CLINICAL TRIAL: NCT01136811
Title: Safety and Efficacy of Computer Assisted Surgery for Use in Vascular Surgery Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated. P.I. left the institution before completing study
Sponsor: University of Chicago (Other)
Collaborators: Louis A. Weiss Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17002A
Record Dates: First submitted 2010-05-28; First posted 2010-06-03 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Lower Extremity Occlusive Disease
MeSH Terms: interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Computer assisted surgery (Experimental)
  Interventions: Device: Computer assisted surgery

INTERVENTIONS:
Device: Computer assisted surgery — use of computer assisted surgical device in vascular surgery
  completion of the proximal (femoral) anastomosis portion of a lower extremity bypass procedure
  Other Names: DaVinci Surgical System

SUMMARY:
The purpose of this study is to evaluate the preliminary safety and efficacy of the daVinci surgical system (computer-assisted surgery) for use in vascular surgery procedures. Although the daVinci Surgical System is FDA approved and widely used for surgical procedures for urology, cardiac, general, and gynecologic procedures, it is not currently approved specifically for use in vascular surgery and the FDA has required the PI to conduct a small feasibility study under an IDE. The investigators are seeking approval by the FDA to utilize the daVinci Surgical System in vascular surgery and to conduct a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant femoropopliteal or tibial occlusive disease not amenable to catheter directed therapy (ie angioplasty/stenting). Symptoms include lifestyle-limiting claudication, rest pain and/or tissue loss.
* Patients with an ABI between 0.2 and 0.8.
* Femoropopliteal disease visible on color duplex ultrasound (DUS)
* Patent and minimally diseased common femoral and proximal superficial artery
* Patients with American Society of Anesthesiology (ASA) I, II or III classification
* PT/PTT, EKG, HbA1c, liver function, within normal ranges within 30 days prior to procedure or stable over the last 6 months.

Current University of Chicago Medical Center Lab standards will be used. Pulmonary function will be assessed as needed by preoperative anesthesia evaluation. (Generally for infrainguinal procedures, pulmonary function is not assessed)

* Body Mass Index (BMI) <40

Exclusion Criteria:

* Previous surgery in the inguinal region (ie: prior femoral artery dissection)
* Myocardial infarction (MI) within the last 6 months
* Laboratory evidence of hypercoagulable state and/or connective tissue disease
* Pregnant women
* History of non-compliance with medical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Chicago, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computer Assisted Surgery
Started | 11
Completed | 0
Not Completed | 11
Not completed — Physician Decision | 11

BASELINE CHARACTERISTICS:
Population: This is to verify that all efforts have been done to contact the PI, however the PI has left the institution since 2011. No one associated with this study works at the institution currently. The current department staff have no access to the data.
  Per IRB records, no analysis was done, the trial was terminated by Principal Investigator and the Principal Investigator has left the institute.
Arm/Group | Computer Assisted Surgery
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: Trial terminated by Principal Investigator and the Principal Investigator has left the institution.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The PI has left the institution since 2011. No one associated with this study works at the institution currently. The current department staff have no access to the data.
  Per IRB records, no analysis was done, the trial was terminated by Principal Investigator and the Principal Investigator has left the institute.
  All efforts have been done to contact the PI and to gather data.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Trial terminated by Principal Investigator and the Principal Investigator has left the institution.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Patency of Graft Anastomosis
Time Frame: 30 Day
Population: The PI has left the institution since 2011. No one associated with this study works at the institution currently. The current department staff have no access to the data.
  Per IRB records, no analysis was done, the trial was terminated by Principal Investigator and the Principal Investigator has left the institute.
  All efforts have been done to contact the PI and to gather data.
Arm/Group | Computer Assisted Surgery
Number analyzed (Participants) | 0

2. Secondary Outcome: Time for Femoral Artery Dissection and Anastomosis
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | Computer Assisted Surgery
Number analyzed (Participants) | 0

3. Secondary Outcome: Improvement in ABI Measurement of 0.15 or Better
Time Frame: 3 month, 6 month, 1 year
Population: as for outcome 1
Arm/Group | Computer Assisted Surgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Death
Description: death
Time Frame: 30day, 1 year
Population: as for outcome 1
Arm/Group | Computer Assisted Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The PI has left the institution since 2011. No one associated with this study works at the institution currently. The current department staff have no access to the data. Per IRB records, no analysis was done, the trial was terminated by Principal Investigator and the Principal Investigator has left the institute. All efforts have been done to contact the PI and to gather data.
Description: The PI has left the institution since 2011. No one associated with this study works at the institution currently. The current department staff have no access to the data.
  Per IRB records, no analysis was done, the trial was terminated by Principal Investigator and the Principal Investigator has left the institute.
  All efforts have been done to contact the PI and to gather data.
Arm/Group | Computer Assisted Surgery
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No